CLINICAL TRIAL: NCT03696563
Title: Automated Administration of Oxygen Using the FreeO2 Device in Ambulances for COPD and Trauma Patients: A Feasibility Study
Brief Title: FreeO2 PreHospital - Automated Oxygen Titration vs Manual Titration According to the BLS-PCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: François Lellouche (Other)
Collaborators: The Ottawa Hospital (Other); Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, François Lellouche, Sponsor, Laval University
Organization: Laval University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20180570-01H
Record Dates: First submitted 2017-12-18; First posted 2018-10-04 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: COPD Exacerbation; Trauma
Keywords: prehospital; oxygen therapy; automation; trauma; COPD
MeSH Terms: conditions — Wounds and Injuries; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This will be a single centered prehospital multi-period cluster crossover feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): In this group, the - usual care based upon BLS-PCS with manual titration of oxygen. In this group the SpO2 was recorded any time with FreeO2 device - recording mode.
  Interventions: Other: Standard administration of oxygen flow
- FreeO2 group (Experimental): The adjustment of the oxygen flow will be made by the FreeO2 system, an automated titration to reach the SpO2 target set by paramedic.
  Interventions: Device: Automated oxygen administration - FreeO2

INTERVENTIONS:
Device: Automated oxygen administration - FreeO2 — The adjustment of the oxygen flow will be made by the FreeO2 system, an automated titration of oxygen flow every second to reach the SpO2 target. The SpO2 target will be set at 90% in COPD patients and 94% in trauma patients.
  Arms: FreeO2 group
Other: Standard administration of oxygen flow — The flow of oxygen will be administered according to the usual protocol during the transport and until transfer to the emergency departement.
  Arms: Control group

SUMMARY:
Evaluation of automated oxygen titration in comparison with manual adjustment oxygen in the out-of-hospital setting by paramedics.

DETAILED DESCRIPTION:
It is a single center study in Ottawa, Ontario Canada.

This will be a single centered prehospital multi-period cluster crossover feasibility trial, enrolling patients in Ottawa, Ontario, who are treated by paramedics from the Ottawa Paramedic Service, who have been trained in the use of the automated oxygen delivery device. We will be using the FreeO2 device. Patients requiring oxygen therapy during prehospital transportation will be enrolled. No randomization will occur within this single centered feasibility study

Patients requiring oxygen therapy during the prehospital transportation will be enrolled and will be included as soon as they are placed into the ambulance, until handover and transfer of care at receiving hospital.

In both groups, SpO2 will be collected continuously every second with FreeO2 monitoring, in addition to the collection of vital signs carried out by the staff according to the standards.

ELIGIBILITY:
Inclusion Criteria:

COPD patient:

1. Known or suspected acute exacerbation of COPD. Acute exacerbation is defined by worsening of the respiratory condition for less than 2 weeks. Suspected COPD is defined by patients of at least 30 years old with respiratory symptoms with a past or current smoking history of at least 10 pack years, or
2. Able to measure SpO2 via pulse oximetry

Trauma patient:

I) Trauma: patients who sustain any trauma (minor or major), II) Able to measure SpO2 via pulse oximetry

Exclusion Criteria:

* Inclusion in another study not allowing the co-enrollment
* Pregnancy
* Age <18 years
* Prehospital Invasive or non-invasive mechanical ventilation
* Meeting high concentration oxygen administration injury or condition (as per BLS-PCS Oxygen Therapy Standard (Version 3.0), s(2)a-f).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the study design - REB approval | Date of REB submission to date of REB approval, target: until 3 months (90 days) from REB submission
  Time to REB approval for single site time to REB approval for single site define by below 3 months (90 days) from REB submission, time to readiness to initiate the clinical trial after REB approval - below 3 months (90 days) from REB approval, evaluation of data collection tool - 100% of data captured in >90% case at hospital discharge (until day 28), Survey responses from Paramedics - At the end of the transportation day
Feasibility of the study design - initiate the clinical trial | Target until 3 months (90 days) from REB approval
  Time to readiness to initiate the clinical trial
Feasibility of the study design - Evaluation of data collection tool | through study completion, an average of 1 year
  target: 100% of data captured in >90% cases
Feasibility of the study design - study protocol compliance | through study completion,an average of 1 year
  Target of 80% of compliance for protocol intervention/control group
Feasibility of the study design - Paramedics survey | through study completion, an average of 1 year
  A survey will be complete by Paramedics at the end of day of transportation (day 1); the target response rate is 75% of case.

SECONDARY OUTCOMES:
Oxygenation - Total Time in the target zone SpO2 | Day 1 - During prehospital transportation (from entry in the ambulance until exit of the ambulance)
  Percentage of time spent in the target zone SpO2
  * 90±2% in the COPD population (in the range of 88 to 92%)
  * 94±2% in the trauma population (in the range of 92 to 96%)
Oxygenation - Total time with hyperoxia | Day 1 - During prehospital transportation (from entry in the ambulance until exit of the ambulance)
  Percentage of time spent in hyperoxia (SpO2 > 94% in COPD patients and SpO2 >98% in trauma patients)
Oxygenation - Total time with hypoxemia | Day 1 - During prehospital transportation (from entry in the ambulance until exit of the ambulance)
  Percentage of time spent in the target zone SpO2
  - % of time with hypoxemia (SpO2<86% in COPD patients and SpO2 <90% in trauma patients)
The oxygentherapy complication- PaCO2 | Day 1- On The first ABG or capillary blood gases after hospital admission
  -Evaluation of level of PaCO2 on the first ABG at ED or ICU admission (when available)
The oxygentherapy complication - respiratory acidosis | Day 1- On The first ABG or capillary blood gases after hospital admission
  -Evaluation of the rate of respiratory acidosis (pH<7.35 and PaCO2>45mmHg) after hospital admission
The rate of patients without oxygen at the end of the transportation | Day 1 - At the end of the transportation (at the exit from the ambulance)
  Rate of patient weaned of oxygen at the end of the transportation
Outcome data - NIV | through study completion, an average of 1 year
  The rate of NIV use during lenght of stay in hospital
Outcome data - ICU admission | through study completion, an average of 1 year
  The rate of ICU admission during lenght of stay in hospital
Outcome data - Death | During hospital stay - hospital admission through study completion or until death if occured, up to 8 weeks
  The rate of death during lenght of stay in hospital
Outcome data | Length of hospital stay measured in calendar days, hospital admission through study completion, up to 8 weeks
  Duration of the hospital length of stay
The oxygen consumption during the pre-hospital transport | Day 1 - During prehospital transportation (from entry in the ambulance until exit of the ambulance),
  Mean O2 flow rate (total O2 consumption) during transportation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Austin, Principal Investigator — Regional Paramedic Program for Eastern Ontario, Ottawa Hospital Research Institute

IPD SHARING:
Plan to Share IPD: No
There is not plan to share individual participant data. All data if shared with be de-identified. Data will be stored on a secure server with access only by study personal.

REFERENCES:
- [Background] Johannigman JA, Branson R, Lecroy D, Beck G. Autonomous control of inspired oxygen concentration during mechanical ventilation of the critically injured trauma patient. J Trauma. 2009 Feb;66(2):386-92. doi: 10.1097/TA.0b013e318197a4bb. PMID 19204511
- [Background] Johannigman JA, Muskat P, Barnes S, Davis K Jr, Beck G, Branson RD. Autonomous control of oxygenation. J Trauma. 2008 Apr;64(4 Suppl):S295-301. doi: 10.1097/TA.0b013e31816bce54. No abstract available. PMID 18385582
- [Background] Higuchi S, Fukushi G, Baba T, Sasaki D, Yoshida Y. New method of testing for carbohydrate absorption in man. Xylose and sucrose absorption; effects of sucrase inhibition. Dig Dis Sci. 1986 Apr;31(4):369-75. doi: 10.1007/BF01311671. PMID 3956333
- [Background] O'Driscoll BR, Howard LS, Davison AG; British Thoracic Society. BTS guideline for emergency oxygen use in adult patients. Thorax. 2008 Oct;63 Suppl 6:vi1-68. doi: 10.1136/thx.2008.102947. No abstract available. PMID 18838559
- [Background] Branson RD, Johannigman JA. Pre-hospital oxygen therapy. Respir Care. 2013 Jan;58(1):86-97. doi: 10.4187/respcare.02251. PMID 23271821
- [Background] Hale KE, Gavin C, O'Driscoll BR. Audit of oxygen use in emergency ambulances and in a hospital emergency department. Emerg Med J. 2008 Nov;25(11):773-6. doi: 10.1136/emj.2008.059287. PMID 18955625
- [Background] Aubier M, Murciano D, Fournier M, Milic-Emili J, Pariente R, Derenne JP. Central respiratory drive in acute respiratory failure of patients with chronic obstructive pulmonary disease. Am Rev Respir Dis. 1980 Aug;122(2):191-9. doi: 10.1164/arrd.1980.122.2.191. PMID 6774639
- [Background] Aubier M, Murciano D, Milic-Emili J, Touaty E, Daghfous J, Pariente R, Derenne JP. Effects of the administration of O2 on ventilation and blood gases in patients with chronic obstructive pulmonary disease during acute respiratory failure. Am Rev Respir Dis. 1980 Nov;122(5):747-54. doi: 10.1164/arrd.1980.122.5.747. PMID 6778278
- [Background] Dunn WF, Nelson SB, Hubmayr RD. Oxygen-induced hypercarbia in obstructive pulmonary disease. Am Rev Respir Dis. 1991 Sep;144(3 Pt 1):526-30. doi: 10.1164/ajrccm/144.3_Pt_1.526. PMID 1909846
- [Background] Sassoon CS, Hassell KT, Mahutte CK. Hyperoxic-induced hypercapnia in stable chronic obstructive pulmonary disease. Am Rev Respir Dis. 1987 Apr;135(4):907-11. doi: 10.1164/arrd.1987.135.4.907. PMID 3565937
- [Background] DAVIES CE, MACKINNON J. Neurological effects of oxygen in chronic cor pulmonale. Lancet. 1949 Nov 12;2(6585):883-5, illust. doi: 10.1016/s0140-6736(49)91459-2. No abstract available. PMID 15393115
- [Background] Wiener AS, Cioffi AF. A group B analogue of subgroup A 3. Am J Clin Pathol. 1972 Dec;58(6):693-7. doi: 10.1093/ajcp/58.6.693. No abstract available. PMID 4629769
- [Background] Murphy R, Mackway-Jones K, Sammy I, Driscoll P, Gray A, O'Driscoll R, O'Reilly J, Niven R, Bentley A, Brear G, Kishen R. Emergency oxygen therapy for the breathless patient. Guidelines prepared by North West Oxygen Group. Emerg Med J. 2001 Nov;18(6):421-3. doi: 10.1136/emj.18.6.421. No abstract available. PMID 11696486
- [Background] Pauwels RA, Buist AS, Calverley PM, Jenkins CR, Hurd SS; GOLD Scientific Committee. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease. NHLBI/WHO Global Initiative for Chronic Obstructive Lung Disease (GOLD) Workshop summary. Am J Respir Crit Care Med. 2001 Apr;163(5):1256-76. doi: 10.1164/ajrccm.163.5.2101039. No abstract available. PMID 11316667
- [Background] Kettel LJ, Diener CF, Morse JO, Stein HF, Burrows B. Treatment of acute respiratory acidosis in chronic obstructive lung disease. JAMA. 1971 Sep 13;217(11):1503-8. No abstract available. PMID 5109747
- [Background] Warren PM, Flenley DC, Millar JS, Avery A. Respiratory failure revisited: acute exacerbations of chronic bronchitis between 1961-68 and 1970-76. Lancet. 1980 Mar 1;1(8166):467-70. doi: 10.1016/s0140-6736(80)91008-9. PMID 6102193
- [Background] Scales DC, Adhikari NK. Lost in (knowledge) translation: "All breakthrough, no follow through"? Crit Care Med. 2008 May;36(5):1654-5. doi: 10.1097/CCM.0b013e3181701525. No abstract available. PMID 18448924
- [Background] Bateman NT, Leach RM. ABC of oxygen. Acute oxygen therapy. BMJ. 1998 Sep 19;317(7161):798-801. doi: 10.1136/bmj.317.7161.798. No abstract available. PMID 9740573
- [Background] DeWitt DS, Prough DS. Blast-induced brain injury and posttraumatic hypotension and hypoxemia. J Neurotrauma. 2009 Jun;26(6):877-87. doi: 10.1089/neu.2007.0439. PMID 18447627
- [Background] Galatius-Jensen S, Hansen J, Rasmussen V, Bildsoe J, Therboe M, Rosenberg J. Nocturnal hypoxaemia after myocardial infarction: association with nocturnal myocardial ischaemia and arrhythmias. Br Heart J. 1994 Jul;72(1):23-30. doi: 10.1136/hrt.72.1.23. PMID 8068464
- [Background] Farquhar H, Weatherall M, Wijesinghe M, Perrin K, Ranchord A, Simmonds M, Beasley R. Systematic review of studies of the effect of hyperoxia on coronary blood flow. Am Heart J. 2009 Sep;158(3):371-7. doi: 10.1016/j.ahj.2009.05.037. Epub 2009 Jul 15. PMID 19699859
- [Background] Floyd TF, Ratcliffe SJ, Detre JA, Woo YJ, Acker MA, Bavaria JE, Resh BF, Pochettino AA, Eckenhoff RA. Integrity of the cerebral blood-flow response to hyperoxia after cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 2007 Apr;21(2):212-7. doi: 10.1053/j.jvca.2006.02.017. Epub 2006 May 18. PMID 17418734
- [Background] Floyd TF, Clark JM, Gelfand R, Detre JA, Ratcliffe S, Guvakov D, Lambertsen CJ, Eckenhoff RG. Independent cerebral vasoconstrictive effects of hyperoxia and accompanying arterial hypocapnia at 1 ATA. J Appl Physiol (1985). 2003 Dec;95(6):2453-61. doi: 10.1152/japplphysiol.00303.2003. Epub 2003 Aug 22. PMID 12937024
- [Background] Johnston AJ, Steiner LA, Gupta AK, Menon DK. Cerebral oxygen vasoreactivity and cerebral tissue oxygen reactivity. Br J Anaesth. 2003 Jun;90(6):774-86. doi: 10.1093/bja/aeg104. PMID 12765894
- [Background] Ronning OM, Guldvog B. Should stroke victims routinely receive supplemental oxygen? A quasi-randomized controlled trial. Stroke. 1999 Oct;30(10):2033-7. doi: 10.1161/01.str.30.10.2033. PMID 10512903
- [Background] Brenner M, Stein D, Hu P, Kufera J, Wooford M, Scalea T. Association between early hyperoxia and worse outcomes after traumatic brain injury. Arch Surg. 2012 Nov;147(11):1042-6. doi: 10.1001/archsurg.2012.1560. PMID 22801994
- [Background] Rincon F, Kang J, Maltenfort M, Vibbert M, Urtecho J, Athar MK, Jallo J, Pineda CC, Tzeng D, McBride W, Bell R. Association between hyperoxia and mortality after stroke: a multicenter cohort study. Crit Care Med. 2014 Feb;42(2):387-96. doi: 10.1097/CCM.0b013e3182a27732. PMID 24164953
- [Background] Rincon F, Kang J, Vibbert M, Urtecho J, Athar MK, Jallo J. Significance of arterial hyperoxia and relationship with case fatality in traumatic brain injury: a multicentre cohort study. J Neurol Neurosurg Psychiatry. 2014 Jul;85(7):799-805. doi: 10.1136/jnnp-2013-305505. Epub 2013 Jun 21. PMID 23794718
- [Background] Cameron L, Pilcher J, Weatherall M, Beasley R, Perrin K. The risk of serious adverse outcomes associated with hypoxaemia and hyperoxaemia in acute exacerbations of COPD. Postgrad Med J. 2012 Dec;88(1046):684-9. doi: 10.1136/postgradmedj-2012-130809. Epub 2012 Sep 12. PMID 22977283
- [Result] Lellouche F, Bouchard PA, Simard S, L'Her E, Wysocki M. Evaluation of fully automated ventilation: a randomized controlled study in post-cardiac surgery patients. Intensive Care Med. 2013 Mar;39(3):463-71. doi: 10.1007/s00134-012-2799-2. Epub 2013 Jan 22. PMID 23338569
- [Result] Lellouche F, Mancebo J, Jolliet P, Roeseler J, Schortgen F, Dojat M, Cabello B, Bouadma L, Rodriguez P, Maggiore S, Reynaert M, Mersmann S, Brochard L. A multicenter randomized trial of computer-driven protocolized weaning from mechanical ventilation. Am J Respir Crit Care Med. 2006 Oct 15;174(8):894-900. doi: 10.1164/rccm.200511-1780OC. Epub 2006 Jul 13. PMID 16840741
- [Result] Denniston AK, O'Brien C, Stableforth D. The use of oxygen in acute exacerbations of chronic obstructive pulmonary disease: a prospective audit of pre-hospital and hospital emergency management. Clin Med (Lond). 2002 Sep-Oct;2(5):449-51. doi: 10.7861/clinmedicine.2-5-449. PMID 12448594
- [Result] Joosten SA, Koh MS, Bu X, Smallwood D, Irving LB. The effects of oxygen therapy in patients presenting to an emergency department with exacerbation of chronic obstructive pulmonary disease. Med J Aust. 2007 Mar 5;186(5):235-8. doi: 10.5694/j.1326-5377.2007.tb00879.x. PMID 17391084
- [Result] Plant PK, Owen JL, Elliott MW. One year period prevalence study of respiratory acidosis in acute exacerbations of COPD: implications for the provision of non-invasive ventilation and oxygen administration. Thorax. 2000 Jul;55(7):550-4. doi: 10.1136/thorax.55.7.550. PMID 10856313
- [Result] Austin MA, Wills KE, Blizzard L, Walters EH, Wood-Baker R. Effect of high flow oxygen on mortality in chronic obstructive pulmonary disease patients in prehospital setting: randomised controlled trial. BMJ. 2010 Oct 18;341:c5462. doi: 10.1136/bmj.c5462. PMID 20959284
- [Result] Wijesinghe M, Perrin K, Ranchord A, Simmonds M, Weatherall M, Beasley R. Routine use of oxygen in the treatment of myocardial infarction: systematic review. Heart. 2009 Mar;95(3):198-202. doi: 10.1136/hrt.2008.148742. Epub 2008 Aug 15. PMID 18708420
- [Result] Lellouche F, L'her E. Automated oxygen flow titration to maintain constant oxygenation. Respir Care. 2012 Aug;57(8):1254-62. doi: 10.4187/respcare.01343. Epub 2012 Feb 17. PMID 22348812